CLINICAL TRIAL: NCT06052436
Title: Open Phase I/IIa Clinical Trial to Evaluate the Safety and Efficacy of Allogenic Administration of Treg Cells Obtained From Thymic Tissue (thyTreg) to Control The Immune Hyperactivation Associated With COVID-19 and/or Acute Respiratory Distress Syndrome
Brief Title: Cell Therapy With Treg Cells Obtained From Thymic Tissue (thyTreg) to Control the Immune Hyperactivation Associated With COVID-19 and/or Acute Respiratory Distress Syndrome (THYTECH2)
Acronym: THYTECH2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Rafael Correa-Rocha, Principal Investigator, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FIBHGM-ECNC003-2021; 2024-519799-25 (EudraCT Number); 2021-003240-25 (Other: AEMPS)
Record Dates: First submitted 2023-09-12; First posted 2023-09-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Immune Hyperactivation; Regulatory T cell; ARDS; COVID-19; Advanced therapy; Immunotherapy; Th1-Th2 Balance
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase A: 5.000.000 thyTreg /kg (Experimental): Allogeneic thyTreg 5.000.000
  Interventions: Biological: Allogeneic thyTreg 5.000.000
- Phase A: standard of care (No Intervention): Standard of care
- Phase B: 10.000.000 thyTreg /kg (Experimental): Allogeneic thyTreg 10.000.000
  Interventions: Biological: Allogeneic thyTreg 10.000.000
- Phase B: standard of care (No Intervention): Standard of care

INTERVENTIONS:
Biological: Allogeneic thyTreg 5.000.000 — Treg lymphocytic cells, differentiated, allogeneic, of thymic tissue, expanded and stimulated with Interleukin (IL-) 2 (thyTreg)
  Other Names: Allogeneic thyTreg cells
  Arms: Phase A: 5.000.000 thyTreg /kg
Biological: Allogeneic thyTreg 10.000.000 — Treg lymphocytic cells, differentiated, allogeneic, of thymic tissue, expanded and stimulated with Interleukin (IL-) 2 (thyTreg)
  Other Names: Allogeneic thyTreg cells
  Arms: Phase B: 10.000.000 thyTreg /kg

SUMMARY:
The investigators developed a GMP protocol to isolate Treg cells from thymic tissue (thyTreg). The thyTreg cells are being evaluated in a Phase I/II clinical trial to evaluate the safety and efficacy of the adoptive transfer of autologous thyTreg to prevent rejection in heart transplant children (NCT04924491), with preliminary results indicating the feasibility and safety of the therapy.

In addition, thyTreg cells have shown low immunogenicity in the pre-clinical setting, indicating that allogeneic use of these thyTreg cells (allo-thyTreg) would have a low risk of adverse effects. These thyTreg cells could inhibit an excessive inflammation in SARS-CoV-2 infection, or ameliorate the immunological affection underlying Acute respiratory distress syndrome, improving life-threatening manifestations, restoring immune balance, and protecting affected tissues.

This clinical trial is an open-label Sequential Parallel Group Phase I/II study to evaluate the safety and efficacy of allogeneic thymus derived Tregs (thyTreg) (thyTreg) in controlling the immune dysregulation associated with SARS-CoV-2 infection and/or Acute Respiratory Distress Syndrome.

DETAILED DESCRIPTION:
The immune system is the body's defense system against pathogens and other harmful agents, but it is also responsible for transplant rejection or autoimmune diseases. Another scenario of disproportionate immune response is the Immune Hyperactivation, an exaggerated systemic inflammatory response such as that caused by respiratory infections like COVID-19, a major cause of acute respiratory distress syndrome (ARDS) in critically ill patients.

The standard treatment to prevent these immune responses is the use of immunosuppressive and immunomodulatory therapy, which produces a pleotropic inhibition on the immune system and have a high cost. However, a widespread feeling among the scientific community is that only re-educating immune system to promote immune tolerance will decline the harmful immune responses without prejudice to the functional integrity of the immune system.

In the context of severe COVID-19 and ARDS, it has been shown that an alteration in the frequency and functionality of Tregs. In addition, it has been described that the increased oxygen therapy requirements is not due to the viral effect, but to the triggered immune hyperinflammation that can lead to multi-organ failure and death. Therefore, although the adoptive transfer of Treg is a promising cell therapy for the treatment of this type of disease, the characteristics of the patients make it unfeasible to obtain enough Treg from the patient to produce a therapeutic dose and, if achieved, the quality of these cells does not allow a prolonged therapeutic effect to be obtained over time.

Tregs are a subset of CD4+ T cells with suppressive function that maintain the immune system balance. Adoptive Treg cell therapy has shown efficacy in a variety of immune-mediated diseases in preclinical and clinical studies. To date, most of the clinical trials employing Treg cell therapy have been limited due to a small Treg numbers obtained (Treg cells represent less than 10% of CD4+ T cells) and the low quality of infused Treg (in terms of purity, survival, and suppressor capacity).

The investigators have developed an innovative Treg manufacturing protocol, that overcome the existing difficulties by employing a new source of cells, which is the thymic tissue routinely removed and discarded in paediatric cardiac surgeries. The protocol allows to produce massive amounts of thymus derived Treg cells (thyTreg), with improved survival, high suppressive capacity and suitable for therapeutic use.

The study will evaluate escalating doses of thyTreg administrated as a single IV dose. The study will include up to 2 cohorts of 4 to 8 subjects per each arm (control group and thyTreg group) followed for a total of 24 months. All subjects will receive standard of care treatment for COVID-19 or ARDS, including dexamethasone and other approved therapies from institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 to 65 years of age
2. Patient Informed and non-opposed to the research by his medical doctor during hospitalization
3. Patient with clinical, radiological, gasometric and immunological criteria defined as:

   1. Acute respiratory failure secondary to acute lung injury of noncardiogenic cause
   2. Pulmonary abnormalities compatible with bilateral alveoloinsterstitial infiltrates by chest imaging (radiograph or scan)
   3. PaO2/FiO2≤ 300 Presence of at least one of the following markers of inflammation: IL6 > 40 pg/ml or ferritin >300 ng/ml or CRP >3 mg/dl or increasing over the last 24 hours

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Body mass index >35
3. Patients not expected to survive 48 hours after enrolment based on clinical assessment
4. Patients with an extracorporeal respiratory support
5. Neutropenia (absolute neutrophil count <1000/uL)
6. Thrombocytopenia (absolute neutrophil count <50000/uL)
7. Positive serology for HBV, HCV, or HIV at Screening
8. Life expectancy of less than 6 months due to other pathologies
9. History of significant underlying pulmonary disease requiring oxygen therapy prior to inclusion.
10. Patients with a history of autoimmune diseases
11. Patients with a history of hematopoietic neoplasia or oncology disease
12. Patients with a history of hematopoietic or solid organ transplant
13. Patients with a congenital or induced immunodeficiency
14. Patients received thymoglobulin, basiliximab or any anti-T-cell therapies within 6 moths prior to the screening visit
15. Patients received other cell therapy in the last 12 months
16. Patients received intravenous immunoglobulin (IVIg) within 5 moths prior to the screening visit
17. Patients who have participated or is participating in a clinical research study evaluating COVID-19 or ARDS within 30 days prior to the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of infusion-related adverse events (safety) by type, frequency, severity, and causality | 24 months

SECONDARY OUTCOMES:
Length of intensive care unit stay | 24 months
Oxygenation improvement as assessed using PaO2/FiO2 and/or SaO2/FiO2 | 24 months
Change in clinical status as assessed using Sequential Organ Failure Assessment Score | 24 months
Change in clinical status as assessed using Acute Physiology and Chronic Health disease Classification System (APACHE) III | 24 months
Change in clinical status as assessed using Barthel score | 24 months
Change in myocardial function as measured by mitral and tricuspid regurgitation using doppler echocardiography | 24 months
Change in myocardial function as measured by mitral and tissue mitral doppler using doppler echocardiography | 24 months
Change in myocardial function as measured by tricuspid and tissue tricuspid using doppler echocardiography | 24 months
Change in SARS-CoV-2 positivity or etiology of ARDS assessed using diagnostics test | 24 months
Change From Baseline in ferritin parameter | 24 months
Change From Baseline in interleukin 6 (IL-6) | 24 months
Change From Baseline in C-Reactive Protein (PCR) | 24 months
Change From Baseline in Treg cells number in peripheral blood | 24 months
Number of T cells, B cells, NK cells, monocytes, dendritic cells, and granulocytes in peripheral blood | 24 months
Change From Baseline in cytokines levels of interferon gamma, tumor necrosis factor alpha and interleukins (IL-6 and IL-10). | 24 months
Overall patient survival rate at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Correa-Rocha, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Spain